CLINICAL TRIAL: NCT00701337
Title: Effect of 17ß-estradiol on Inflammatory-immune Responses in Post-menopausal Women According to Administration Route: Pilot Study
Brief Title: Effect of 17ß-estradiol on Inflammatory-immune Responses in Post-menopausal Women According to Administration Route
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0507402
Record Dates: First submitted 2007-02-22; First posted 2008-06-19 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Postmenopausal
Keywords: Estrogen Replacement Therapy; menopausal women
MeSH Terms: interventions — Estradiol; estradiol, estriol drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 Oral (Experimental): oestradiol by oral administration - Estrofem 2 mg
  Interventions: Drug: oestradiol
- 2 patch (Experimental): oestradiol par patch - Estrapatch 60microg/24h
  Interventions: Drug: oestradiol

INTERVENTIONS:
Drug: oestradiol — oestradiol 2 mg oral route 30 days
  Other Names: Estrofem
  Arms: 1 Oral
Drug: oestradiol — oestradio transdermal patch 60ug by 24 hours 30 days
  Other Names: Oestrapatch
  Arms: 2 patch

SUMMARY:
The aim of this pilot study conducted in post-menopausal women is to evaluate the effect of 17ß-estradiol administration on inflammatory-immune cells, namely antigen-presenting cells (monocytes/dendritic cells), and more precisely on their activation by inflammatory stimuli. This study will allow us to determine our ability to recruit menopausal women and to characterize the optimal primary end-point among the numerous criteria tested

DETAILED DESCRIPTION:
Although the beneficial effects of hormonal replacement therapy (HRT) against osteoporosis and climacteric symptoms have been clearly established, randomized studies recently revealed that the combined administration of oral estrogens and medroxyprogesterone acetate increases the incidence of coronary events and strokes during the first months of treatment. Furthermore, oral estrogens significantly enhance IL-6 and CRP secretion. This increase in the plasma concentration of inflammatory markers probably results from a direct effect of oral administration on the liver, since i twas not observed with estrogens administered by transdermal route.

Our experimental data in ovariectomized mice demonstrated that the chronic subcutaneous administration of17ß-estradiol (E2) enhances the expression of pro-inflammatory cytokines by Th1 lymphocytes, Natural Killer T cells and monocytes/macrophages. This pro-inflammatory effect of E2 could play a role in the deleterious vascular effects observed in randomized studies, especially by favoring plaque instability.

Our aim is to determine whether E2 administration in menopausal women leads to an inflammatory phenotype of circulating antigen-presenting cells, especially monocytes. Indeed, evaluating the inflammatory status at the cellular level probably gives more precise informations than plasma cytokine concentrations to predict the ability of estrogens to enhance inflammatory processes. We first propose a pilot study in order to determine enrollment feasibility, as well as the optimal biological endpoints to assess monocyte activation status. These latter criteria will be then used in a future randomized study comparing two routes of E2 administration (oral vs transdermal).

The present study will include 34 menopausal women. After the inclusion visit, three visits will be performed with the collection of a 50 ml blood sample and the isolation of circulating immune cells (monocytes).

The following criteria will be studied before (V1 and V2) and after 30 ± 3 days of E2 treatment (V3:

1. expression of surface activation molecules.
2. Secretion of cytokines in response to several Toll-like receptor stimuli.
3. IL-6 and CRP-US plasma concentrations.

We will first assess the intra-individual variability (V1 and V2). At visit 2 (V2), the subjects will be randomized to receive E2 either by oral (n= 17) or transdermal (n= 17) route.

ELIGIBILITY:
Inclusion Criteria:

* Women with confirmed menopause (duration : 1 to 5 years)
* No contra-indication of hormonal replacement therapy due to medical history
* Mammogram without significant abnormality (< 12 months)
* Normal body mass index (BMI) (19 ≤ IMC ≤ 25 kg/m2)
* No treatment with estrogens and/or progestatives and/or SERM (specific moduator of estrogen receptor) and/or phytoestrogènes ongoing or stopped for less than 3 months
* No clinical or biological abnormality or treatment indicating the presence of an infectious or inflammatory disease.
* No participation to another clinical study during the 3 months before the inclusion
* Ability to sign the consent form.

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2006-09; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
To determine the feasibility of a future multicentric randomized trial : estimation of the number of subjects required | 1 month

SECONDARY OUTCOMES:
variability and repeatability of the biological parameters studied | 1 month
  number of circulating immune cells, expression of surface molecules by monocytes, secretion of cytokines following TLR activation
Feasibility of the recruitment, enrollment and follow-up of menopausal women | End of study

CONTACTS AND LOCATIONS:
Overall Officials: Pierre GOURDY, Principal Investigator — Hospital University Toulouse
Locations (1):
- University Hospital Toulouse, Toulouse, France

REFERENCES:
- [Result] Seillet C, Laffont S, Tremollieres F, Rouquie N, Ribot C, Arnal JF, Douin-Echinard V, Gourdy P, Guery JC. The TLR-mediated response of plasmacytoid dendritic cells is positively regulated by estradiol in vivo through cell-intrinsic estrogen receptor alpha signaling. Blood. 2012 Jan 12;119(2):454-64. doi: 10.1182/blood-2011-08-371831. Epub 2011 Nov 16. PMID 22096248